CLINICAL TRIAL: NCT06120114
Title: Prospective Pilot Trial of Laparoscopic High-Ligation Repair of Indirect Inguinal Hernias in Adults
Brief Title: Laparoscopic High-Ligation Repair of Indirect Inguinal Hernias in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Petter Fosse Gjessing, MD,PhD, Consultant Surgeon, University Hospital of North Norway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1053(REK)
Record Dates: First submitted 2023-10-24; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Inguinal Hernia, Indirect; Surgery; Postoperative Pain; Recurrence
Keywords: Laparoscopy; Inguinal; Hernia; Indirect
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Recurrence; Hernia

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified percutaneous internal ring suturing (Experimental): Patients with indirect inguinal hernia operated with modified percutaneous internal ring suturing
  Interventions: Procedure: Modified percutaneous internal ring suturing

INTERVENTIONS:
Procedure: Modified percutaneous internal ring suturing — Laparoscopically guided percutaneous high ligation of indirect inguinal hernia in adults
  Other Names: PIRS

SUMMARY:
Inguinal hernia surgery has undergone significant and extensive transformation, including the advent of tissue-based repairs and later, tension-free repairs with the acceptance of prosthetic mesh. However, there is still significant pain associated with the use of mesh, as well as the risk of potential injury to neurovascular structures. In the pediatric population, non-mesh laparoscopic high-ligation repair of indirect inguinal hernias is one of the most common procedures performed. High-ligation of indirect inguinal hernias in the adolescent population is also effective, with a low recurrence rate and low incidence of chronic symptoms, but this technique is uncommonly used by adult hernia surgeons due to concern for recurrence.The purpose of this study is to conduct a pilot trial to examine the efficacy of high-ligation repair of indirect inguinal hernias in adult patients.

Our hypothesis is that the laparoscopic, non-mesh repair technique is an effective method of repairing indirect inguinal hernias, with an acceptable recurrence rate and decreased postoperative pain. This pilot trial will allow the design of a randomized clinical trial comparing the efficacy of this technique to other standard repair techniques.

DETAILED DESCRIPTION:
Recruitment:

The participants will be recruited from the Department of Digestive Surgery, University Hospital North Norway, Tromsø. The patient will be asked to participate in the study after evaluation by the principal investigator when candidacy has been established. The investigator or study staff will discuss the study with the patient and the study staff will participate in reviewing details and questions regarding the study if necessary. For each subject, written informed consent will be obtained prior to any protocol-related activities. As part of this procedure, the principal investigator or one of the associates must explain orally and in writing the nature, duration, and purpose of the study in such a manner that the subject is aware of the potential risks, inconveniences, or adverse effects that may occur. Patients should be informed that the subject may withdraw from the study at any time.

Preoperative evaluation:

All patients will undergo our standard pre-operative evaluation and at this visit it will be determined if the patient is a candidate for this study. At this study visit, the doctor will ask about past medical and surgical history and any medications the patient is taking and conduct a physical examination. If the patient qualifies for study participation, the patient will be asked to join the study. If the patient chooses to participate, the study staff will collect additional information such as gender, age, height, weight, medical and surgical history, and information relating to the hernia. Patients will be asked to fill out and complete 3 quality of life questionnaires (Short Form-36, Activities Assessment and a Surgical Site Pain Scale) that ask about activities and how the hernia impacts what they can do.

Study intervention:

On the day that the hernia is repaired, the surgery will be performed in the laparoscopic manner, without the use of mesh reinforcement material. As part of the study, the surgeon will collect information about the hernia and surgery, such as the size and length of the hernia, operative time. A 10 mm incision is made below the umbilicus. A 10 mm trocar and camera are inserted through the umbilical incision and the abdomen is insufflated to 12 mm Hg. An extra 5 mm Maryland dissector is inserted through a 5 mm trocar in the lower left quadrant of the abdominal wall. A small 1 mm incision is made in the inguinal area. Hydrodissection with 0.25% bupivacaine is carried out to disassociate the peritoneum from the inguinal canal cord structures. Next, an 19-gauge spinal needle is prepared by threading a loop of 3-0 Prolene suture into the barrel of the needle. The needle is inserted through the inguinal incision and pierces the peritoneum to enter the abdominal cavity. No injury to the cord structures occurs because of the previous hydrodissection technique. The Prolene loop is threaded through the needle, and the needle is pulled out of the abdominal wall, leaving the suture loop in place. A second loop of 3-0 Prolene suture is threaded into a new 19-gauge spinal needle. This second threaded needle is inserted through the same inguinal incision and pierces through the peritoneum at or near the same point of the first needle. The first suture loop is lassoed around the needle, before the second suture loop is threaded out of the needle and into the abdominal cavity. The needle is pulled out, leaving both suture loops in the abdominal cavity, with the first loop threaded around the second loop. Next, the first suture loop is pulled out of the abdominal wall, which snares the second loop along with it and closes the inguinal hernia defect as it pulls through. The Prolene suture is then exchanged with a braided 2-0 Ethibond (non-absorbable) suture by pulling through the incision site. This suture is doubly ligated. After desufflation of the abdominal cavity, the fascia below the umbilicus and the skin incisions are closed with sutures. The operative time is predicted to be between 20-60 minutes.

Follow-up:

Patients will be given instructions to return to the surgeon's clinic to be examined by their surgeon at 1 month (+/- 2 weeks), and 1 year (+/- 1 month) following surgery. The patients will have their abdominal wound evaluated and be examined for general health and hernia recurrence. They will be asked about any medications they are taking and about any problems they may have had with their hernia repair. Information about any procedures that may be performed during this time will be collected. Patients will be asked to complete the same surveys that they filled out prior to surgery at each of these visits. If at any time throughout the study a hernia recurrence is suspected clinically, then a physical examination will be performed to evaluate the repair.

Data confidentiality:

All information collected, such as name or medical record number will be in a password/firewall protected computer to which only the investigators will have access. All research data will be recorded and stored in a locked office in the Department of Digestive Surgery. All Photographs will be stored separately in a locked cabinet and de-identified by a subject identification number. Only investigators and members of the research team will have key access.

Data analysis:

Since this is a pilot trial, there is no comparison or control arm in this study. Statistical tests will be used when appropriate, but otherwise the purpose of this study will be to report outcomes and feasibility.

Research related injury:

If injury occurs as a result of the involvement in this research, medical treatment will be given by, or under the auspices of the Dept of Digestive Surgery.

ELIGIBILITY:
Inclusion Criteria:

• Subjects who present to the office of the study investigators for repair of an indirect inguinal hernia

Exclusion Criteria:

* Recurrent hernia
* Emergent cases
* Cirrhosis or liver disease (bilirubin > 3 mg/dL).
* Subjects on dialysis
* Subjects with collagen vascular disease
* BMI over 35 kg/m2
* Bilateral inguinal hernias
* Direct inguinal hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-20 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2023-10-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with inguinal hernia recurrence | One month and one year after surgery
  Number of patients with recurrence determined by clinical examination

SECONDARY OUTCOMES:
Degree of pain related to the hernia or hernia surgery | Prior to surgery and one month and one year after surgery
  Four 150 mm visual analog surgical pain scales (Scores 0-150, higher score = worse outcome)
Health related quality of life | Prior to surgery and one month and one year after surgery
  36-Item Short Form Health Survey (Scores 0-100, higher score = better outcome
physical activity levels assessed by scale | Prior to surgery and one month and one year after surgery
  Activities Assessment Scale (Scores 0-100, higher score = better outcome)

OTHER OUTCOMES:
Number of patients with self-reported inguinal hernia recurrence | Through study completion, a median of 89 months
  Number of patients with self-reported recurrence by telephone interview

CONTACTS AND LOCATIONS:
Overall Officials: Rolv-Ole Lindsetmo, Principal Investigator — University Hospital North Norway

IPD SHARING:
Plan to Share IPD: No